CLINICAL TRIAL: NCT01584648
Title: A Phase III, Randomized, Double-blinded Study Comparing the Combination of the BRAF Inhibitor, Dabrafenib and the MEK Inhibitor, Trametinib to Dabrafenib and Placebo as First-line Therapy in Subjects With Unresectable (Stage IIIC) or Metastatic (Stage IV) BRAF V600E/K Mutation-positive Cutaneous Melanoma
Brief Title: A Study Comparing Trametinib and Dabrafenib Combination Therapy to Dabrafenib Monotherapy in Subjects With BRAF-mutant Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115306; 2011-006087-49 (EudraCT Number); CDRB436B2301 (Other: Novartis)
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Melanoma
Keywords: Randomized study; combination therapy; BRAF inhibitor; GSK1120212; BRAF V600E/K mutation-positive cutaneous melanoma; trametinib; GSK2118436; MEK inhibitor; Phase III; dabrafenib
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dabrafenib + Trametinib (Experimental): Dabrafenib and Trametinib combination
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Dabrafenib + Placebo (Active Comparator): Dabrafenib and Trametinib placebo
  Interventions: Drug: Dabrafenib; Drug: Trametinib placebo

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib 150 mg twice daily
  Other Names: GSK2118436
Drug: Trametinib — Trametinib 2 mg once daily
  Other Names: GSK1120212
  Arms: Dabrafenib + Trametinib
Drug: Trametinib placebo — Dabrafenib 150 mg twice daily and trametinib placebo
  Other Names: Placebo
  Arms: Dabrafenib + Placebo

SUMMARY:
This was a two-arm, double-blinded, randomized, Phase III study comparing dabrafenib and trametinib combination therapy to dabrafenib administered with a placebo (dabrafenib monotherapy). Subjects with histologically confirmed cutaneous melanoma that is either Stage IIIC (unresectable) or Stage IV, and BRAF V600E/K mutation positive were screened for eligibility. Subjects who had prior systemic anti-cancer treatment in the advanced or metastatic setting were not eligible although prior systemic treatment in the adjuvant setting was allowed. Subjects were stratified according to the baseline lactate dehydrogenase level and BRAF genotype.

DETAILED DESCRIPTION:
Dabrafenib and trametinib was administered orally at their recommended monotherapy doses of 150 mg b.i.d and 2 mg q.d., respectively. Subjects in the combination therapy arm received both agents; subjects in the dabrafenib monotherapy arm received dabrafenib and placebo. Treatment was continued in both arms until disease progression, death, unacceptable toxicity, or withdrawal of consent.

After treatment discontinuation, subjects were followed for survival and disease progression as applicable to collect data for the secondary objective of overall survival (OS).

Crossover to the combination therapy arm was allowed for subjects still receiving study treatment on the dabrafenib monotherapy arm after the positive result for the final OS analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cutaneous melanoma that is either Stage IIIC (unresectable) or Stage IV (metastatic), and determined to be BRAF V600E/K mutation-positive using the bioMerieux (bMx) investigational use only (IUO) THxID BRAF Assay (IDE: G120011). The assay will be conducted by a central reference laboratory. Subjects with ocular or mucosal melanoma are not eligible.
* The subject must have a radiologically measurable tumor
* The subject is able to carry out daily life activities without significant difficulty (ECOG performance status score of 0 or 1).
* Able to swallow and retain oral medication
* Sexually active subjects must use acceptable methods of contraception during the course of the study
* Adequate organ system function and blood counts

Exclusion Criteria:

* Prior treatment with a BRAF or a MEK inhibitor
* Prior systemic anti-cancer treatment for Stage IIIC (unresectable) or Stage IV (metastatic) melanoma. Prior systemic treatment in the adjuvant setting is allowed. (Note: Ipilimumab treatment must end at least 8 weeks prior to randomization.)
* The subject has received major surgery or certain tyes of cancer therapy with 21 days of starting treatment
* Current use of prohibited medication listed in the protocol
* Left ventricular ejection fraction less than the lower limit of normal
* Uncontrolled blood pressurl
* History or current evidence of retinal vein occlusion or central serous retinopathy
* Brain metastases unless previously treated with surgery or stereotactic radiosurgery and the disease has been stable for at least 12 weeks
* The subject is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2012-05-04 (Actual); Primary Completion 2013-08-26 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (108):
- United States (18):
  - Novartis Investigative Site, Scottsdale, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Columbia, South Carolina
  - Novartis Investigative Site, Chattanooga, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Richmond, Virginia
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
- Australia (6):
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Canada (5):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (7):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (29):
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Heilbronn, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg, Bavaria
  - Novartis Investigative Site, Erlangen, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Darmstadt, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Buxtehude, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Homburg, Saarland
  - Novartis Investigative Site, Dresden, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Erfurt, Thuringia
  - Novartis Investigative Site, Gera, Thuringia
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Berlin
- Greece (3):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, N. Faliro
  - Novartis Investigative Site, Thessaloniki
- Italy (6):
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Bergamo, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Candiolo (TO), Piedmont
  - Novartis Investigative Site, Padua, Veneto
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Zwolle
- Russia (4):
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Spain (4):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Valencia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Ukraine (6):
  - Novartis Investigative Site, Dnipropetrovsk
  - Novartis Investigative Site, Donetsk
  - Novartis Investigative Site, Khmelnytskyi
  - Novartis Investigative Site, Kyiv
  - Novartis Investigative Site, Lviv
  - Novartis Investigative Site, Sumy
- United Kingdom (11):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Aberdeen
  - Novartis Investigative Site, Bebington
  - Novartis Investigative Site, Edgbaston, Birmingham
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Preston

REFERENCES:
- [Derived] Schadendorf D, Robert C, Dummer R, Flaherty KT, Tawbi HA, Menzies AM, Banerjee H, Lau M, Long GV. Pyrexia in patients treated with dabrafenib plus trametinib across clinical trials in BRAF-mutant cancers. Eur J Cancer. 2021 Aug;153:234-241. doi: 10.1016/j.ejca.2021.05.005. Epub 2021 Jul 2. PMID 34225229
- [Derived] Syeda MM, Wiggins JM, Corless BC, Long GV, Flaherty KT, Schadendorf D, Nathan PD, Robert C, Ribas A, Davies MA, Grob JJ, Gasal E, Squires M, Marker M, Garrett J, Brase JC, Polsky D. Circulating tumour DNA in patients with advanced melanoma treated with dabrafenib or dabrafenib plus trametinib: a clinical validation study. Lancet Oncol. 2021 Mar;22(3):370-380. doi: 10.1016/S1470-2045(20)30726-9. Epub 2021 Feb 12. PMID 33587894
- [Derived] Robert C, Grob JJ, Stroyakovskiy D, Karaszewska B, Hauschild A, Levchenko E, Chiarion Sileni V, Schachter J, Garbe C, Bondarenko I, Gogas H, Mandala M, Haanen JBAG, Lebbe C, Mackiewicz A, Rutkowski P, Nathan PD, Ribas A, Davies MA, Flaherty KT, Burgess P, Tan M, Gasal E, Voi M, Schadendorf D, Long GV. Five-Year Outcomes with Dabrafenib plus Trametinib in Metastatic Melanoma. N Engl J Med. 2019 Aug 15;381(7):626-636. doi: 10.1056/NEJMoa1904059. Epub 2019 Jun 4. PMID 31166680
- [Derived] Long GV, Grob JJ, Nathan P, Ribas A, Robert C, Schadendorf D, Lane SR, Mak C, Legenne P, Flaherty KT, Davies MA. Factors predictive of response, disease progression, and overall survival after dabrafenib and trametinib combination treatment: a pooled analysis of individual patient data from randomised trials. Lancet Oncol. 2016 Dec;17(12):1743-1754. doi: 10.1016/S1470-2045(16)30578-2. Epub 2016 Nov 16. PMID 27864013
- [Derived] Long GV, Stroyakovskiy D, Gogas H, Levchenko E, de Braud F, Larkin J, Garbe C, Jouary T, Hauschild A, Grob JJ, Chiarion-Sileni V, Lebbe C, Mandala M, Millward M, Arance A, Bondarenko I, Haanen JB, Hansson J, Utikal J, Ferraresi V, Kovalenko N, Mohr P, Probachai V, Schadendorf D, Nathan P, Robert C, Ribas A, DeMarini DJ, Irani JG, Swann S, Legos JJ, Jin F, Mookerjee B, Flaherty K. Dabrafenib and trametinib versus dabrafenib and placebo for Val600 BRAF-mutant melanoma: a multicentre, double-blind, phase 3 randomised controlled trial. Lancet. 2015 Aug 1;386(9992):444-51. doi: 10.1016/S0140-6736(15)60898-4. Epub 2015 May 31. PMID 26037941
- [Derived] Schadendorf D, Amonkar MM, Stroyakovskiy D, Levchenko E, Gogas H, de Braud F, Grob JJ, Bondarenko I, Garbe C, Lebbe C, Larkin J, Chiarion-Sileni V, Millward M, Arance A, Mandala M, Flaherty KT, Nathan P, Ribas A, Robert C, Casey M, DeMarini DJ, Irani JG, Aktan G, Long GV. Health-related quality of life impact in a randomised phase III study of the combination of dabrafenib and trametinib versus dabrafenib monotherapy in patients with BRAF V600 metastatic melanoma. Eur J Cancer. 2015 May;51(7):833-40. doi: 10.1016/j.ejca.2015.03.004. Epub 2015 Mar 17. PMID 25794603
- [Derived] Menzies AM, Ashworth MT, Swann S, Kefford RF, Flaherty K, Weber J, Infante JR, Kim KB, Gonzalez R, Hamid O, Schuchter L, Cebon J, Sosman JA, Little S, Sun P, Aktan G, Ouellet D, Jin F, Long GV, Daud A. Characteristics of pyrexia in BRAFV600E/K metastatic melanoma patients treated with combined dabrafenib and trametinib in a phase I/II clinical trial. Ann Oncol. 2015 Feb;26(2):415-21. doi: 10.1093/annonc/mdu529. Epub 2014 Nov 18. PMID 25411413
- [Derived] Long GV, Stroyakovskiy D, Gogas H, Levchenko E, de Braud F, Larkin J, Garbe C, Jouary T, Hauschild A, Grob JJ, Chiarion Sileni V, Lebbe C, Mandala M, Millward M, Arance A, Bondarenko I, Haanen JB, Hansson J, Utikal J, Ferraresi V, Kovalenko N, Mohr P, Probachai V, Schadendorf D, Nathan P, Robert C, Ribas A, DeMarini DJ, Irani JG, Casey M, Ouellet D, Martin AM, Le N, Patel K, Flaherty K. Combined BRAF and MEK inhibition versus BRAF inhibition alone in melanoma. N Engl J Med. 2014 Nov 13;371(20):1877-88. doi: 10.1056/NEJMoa1406037. Epub 2014 Sep 29. PMID 25265492

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 103 centers in 14 countries worldwide: Argentina (1), Australia (6), Canada (5), France (8), Germany (25), Greece (3), Italy (8), Netherlands (3), Russia (4), Spain (7), Sweden (4), Ukraine (7), United Kingdom (10), and USA (12).
Pre-assignment Details: Approximately, 340 subjects were planned to be randomized in a 1:1 ratio (170 subjects each in combination therapy and monotherapy). A total of 423 subjects with unresectable or metastatic, BRAF V600E or V600K mutation-positive melanoma were randomized to dabrafenib and trametinib (n=211) or dabrafenib and placebo (n=212).
Groups:
- Dabrafenib + Trametinib: Participants received dabrafenib 150 milligram (mg) HPMC capsules orally twice daily (BID), once in the morning and a second dose approximately 12 hours after the morning dose, and trametinib 2 mg once daily in the morning. Treatment was continued until disease progression, death, unacceptable toxicity, or withdrawal of consent.
- Dabrafenib + Placebo: Participants received dabrafenib 150 mg HPMC capsules orally BID, once in the morning and a second dose approximately 12 hours after the morning dose, and trametinib placebo once daily in the morning. Treatment was continued until disease progression, death, unacceptable toxicity, or withdrawal of consent. Crossover to the combination therapy arm was allowed for subjects still receiving study treatment on the dabrafenib monotherapy arm after the positive result for the final OS analysis.
Period: Overall Study
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Started (All randomized patients included into Intent-to-Treat (ITT) population.) | 211 | 212
Safety Set (All patients who received at least one dose of study treatment) | 209 | 211
Crossover Population (All monotherapy randomized patients who crossed over to combination therapy) | 0 | 28
Completed | 0 | 0
Not Completed | 211 | 212
Not completed — Death | 136 | 146
Not completed — Lost to Follow-up | 9 | 9
Not completed — Investigator discretion | 3 | 2
Not completed — Withdrew consent | 13 | 4
Not completed — Study closed/terminated | 50 | 23
Not completed — Crossover to Dabrafenib + Trametinib | 0 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo | Total
Number analyzed (Participants) | 211 | 212 | 423
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (13.33) | 55.3 (13.75) | 55.2 (13.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 98 | 198
  Male | 111 | 114 | 225
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 0 | 1 | 1
  White - White/Caucasian/European Heritage | 211 | 211 | 422

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Investigator
Description: PFS is defined as the interval between the date of randomization and the earliest date of PD or death due to any cause. PD was based on radiographic or photographic evidence, and assessments were made by the investigator according to RECIST, version 1.1. PD is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started. In addition, the sum must have an absolute increase from nadir of 5 mm. The appearance of one or more new lesions, or the worsening of non-target lesions significant enough to require study treatment discontinuation, was also included as PD. Participants who received anti-cancer therapy prior to the date of documented events, were censored at the last adequate assessment prior to the initiation of therapy. If the participant did not have documented progression or death, PFS was censored at the date of the last adequate assessment.
Time Frame: From randomization until the earliest date of disease progression (PD) or death due to any cause (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population was considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Number analyzed (Participants) | 211 | 212
Months | 10.2 [8.1 to 12.8] | 8.8 [5.9 to 9.3]
Statistical Analysis 1: Comparison: Dabrafenib + Trametinib vs Dabrafenib + Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.59 to 0.91] — Hazard ratios (HRs) were estimated using a Pike estimator

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval of time between the date of randomization and the date of death due to any cause. For the participants who did not die, overall survival was censored at the date of last contact.
Time Frame: From the date of randomization until date of death due to any cause (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population was considered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Number analyzed (Participants) | 211 | 212
Months | 25.8 [19.2 to 38.2] | 18.7 [15.2 to 23.1]
Statistical Analysis 1: Comparison: Dabrafenib + Trametinib vs Dabrafenib + Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.64 to 1.02] — Hazard ratios (HRs) were estimated using a Pike estimator

3. Secondary Outcome: Objective Response Rate (ORR) as Assessed by the Investigator
Description: ORR is defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR). A participant was defined as a responder if he/she sustained a complete response (CR: the disappearance of all target lesions and any pathological lymph nodes must have a short axis of <10 mm and the disappearance of all non-target lesions) or partial response (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters or the persistence of 1 or more non-target lesions or lymph nodes identified as a site of disease at Baseline with a short axis of ≥10mm). Only descriptive analysis performed.
Time Frame: From randomization until the first documented complete response or partial response (up to approximately 6 years)
Population: Intent-to-Treat (ITT) Population was considered. Only participants with measurable disease at Baseline per RECIST were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Number analyzed (Participants) | 210 | 210
Participants | 146 | 113

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the first documented complete response (CR: the disappearance of all target lesions and any pathological lymph nodes must have a short axis of <10 mm and the disappearance of all non-target lesions) or partial response (PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the Baseline sum of the diameters or the persistence of 1 or more non-target lesions or lymph nodes identified as a site of disease at Baseline with a short axis of ≥10mm) until disease progression (PD) or death due to any cause. PD is defined as at least a 20% increase in the sum of the diameters of target lesions with an absolute increase of at least 5mm or the appearance of one or more new lesions, or the worsening of non target lesions significant enough to require study treatment discontinuation. PD was based on the radiological evidence by investigator. Only descriptive analysis performed.
Time Frame: From the time of the first documented response (CR or PR) until disease progression (up to approximately 6 years)
Population: ITT population. Only those participants with a confirmed CR or PR were analyzed (with or without measurabe disease at Baseline).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Number analyzed (Participants) | 146 | 114
Months | 12.9 [9.3 to 18.4] | 10.2 [8.3 to 13.8]

5. Secondary Outcome: Trametinib Pharmacokinetic Concentrations
Description: Blood samples were collected for Pharmacokinetic (PK) analysis in all participants. Three blood samples were collected at Week 8: pre-dose, 1-3 hours post dose, and 4-6 hours post dose. One pre-dose blood sample was obtained at Weeks 16 and 24. Only descriptive analysis performed.
Time Frame: Week 8 (0, 1-3, 4-6 hours post dose), Weeks 16 and 24 (0 hour pre-dose)
Population: Pharmacokinetic (PK) Population: all participants included in the safety population for whom a PK sample was obtained and analyzed. Only participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Number analyzed (Participants) | 203 | 194
Nanogram per Milliliter (ng/mL)
  Week 8, pre-dose: number analyzed (Participants) | 176 | 170
  Week 8, pre-dose | 9.9209 (3.86587) | 0.0000 (0.00000)
  Week 8, 1-3 hours: number analyzed (Participants) | 176 | 176
  Week 8, 1-3 hours | 19.0382 (6.86542) | 0.0261 (0.34598)
  Week 8, 4-6 hours: number analyzed (Participants) | 174 | 171
  Week 8, 4-6 hours | 16.7496 (5.64363) | 0.0000 (0.00000)
  Week 16 pre-dose: number analyzed (Participants) | 179 | 162
  Week 16 pre-dose | 11.0385 (4.79185) | 0.0039 (0.03548)
  Week 24 pre-dose: number analyzed (Participants) | 157 | 130
  Week 24 pre-dose | 11.5167 (5.19171) | 0.0548 (0.62447)

6. Secondary Outcome: Dabrafenib and Dabrafenib Metabolites (Hydroxy-, Carboxy- and Desmethyl-Dabrafenib) Concentrations
Description: Blood samples were collected for PK analysis in all participants. Three blood samples were collected at Week 8: pre-dose, 1-3 hours post dose, and 4-6 hours post dose. One pre-dose blood sample was obtained at Weeks 16 and 24. Plasma concentrations of Dabrafenib (GSK2118436) and its metabolites (Hydroxy-Dabrafenib (GSK2285403), Carboxy-Dabrafenib (GSK2298683), and Desmethyl-Dabrafenib (GSK2167542)) were determined using the currently approved analytical methodology. Only descriptive analysis performed.
Time Frame: Week 8 (0, 1-3, 4-6 hours post dose), Weeks 16 and 24 (0 hour pre-dose)
Population: PK Population.
Measure: Mean (Standard Deviation); unit: Nanogram per Milliliter (ng/mL)
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo
Number analyzed (Participants) | 203 | 194
Nanogram per Milliliter (ng/mL)
  GSK2118436, Week 8, pre-dose: number analyzed (Participants) | 176 | 170
  GSK2118436, Week 8, pre-dose | 92.1 (204.85) | 64.4 (96.98)
  GSK2118436, Week 8, 1-3 hours: number analyzed (Participants) | 176 | 176
  GSK2118436, Week 8, 1-3 hours | 1309.6 (982.25) | 1362.3 (992.97)
  GSK2118436, Week 8, 4-6 hours: number analyzed (Participants) | 173 | 171
  GSK2118436, Week 8, 4-6 hours | 458.9 (318.59) | 539.7 (553.09)
  GSK2118436, Week 16 pre-dose: number analyzed (Participants) | 179 | 162
  GSK2118436, Week 16 pre-dose | 151.6 (261.31) | 151.02 (381.32)
  GSK2118436, Week 24 pre-dose: number analyzed (Participants) | 157 | 130
  GSK2118436, Week 24 pre-dose | 167.0 (346.97) | 156.5 (357.50)
  GSK2285403, Week 8, pre-dose: number analyzed (Participants) | 176 | 170
  GSK2285403, Week 8, pre-dose | 346.6 (261.73) | 308.9 (224.56)
  GSK2285403, Week 8, 1-3 hours: number analyzed (Participants) | 176 | 176
  GSK2285403, Week 8, 1-3 hours | 361.7 (245.92) | 341.8 (240.96)
  GSK2285403, Week 8, 4-6 hours: number analyzed (Participants) | 174 | 171
  GSK2285403, Week 8, 4-6 hours | 316.9 (208.51) | 328.1 (234.95)
  GSK2285403, Week 16 pre-dose: number analyzed (Participants) | 179 | 162
  GSK2285403, Week 16 pre-dose | 335.0 (228.26) | 331.0 (250.04)
  GSK2285403, Week 24 pre-dose: number analyzed (Participants) | 157 | 130
  GSK2285403, Week 24 pre-dose | 306.2 (203.77) | 312.8 (250.28)
  GSK2298683, Week 8, pre-dose: number analyzed (Participants) | 176 | 172
  GSK2298683, Week 8, pre-dose | 82.0 (123.93) | 76.7 (109.09)
  GSK2298683,Week 8, 1-3 hours: number analyzed (Participants) | 177 | 179
  GSK2298683,Week 8, 1-3 hours | 648.5 (459.01) | 672.7 (519.45)
  GSK2298683, Week 8, 4-6 hours: number analyzed (Participants) | 174 | 173
  GSK2298683, Week 8, 4-6 hours | 391.3 (206.70) | 502.2 (356.72)
  GSK2298683, Week 16 pre-dose: number analyzed (Participants) | 179 | 163
  GSK2298683, Week 16 pre-dose | 128.7 (174.26) | 121.1 (195.15)
  GSK2298683,Week 24 pre-dose: number analyzed (Participants) | 156 | 130
  GSK2298683,Week 24 pre-dose | 126.1 (219.82) | 145.7 (265.57)
  GSK2167542, Week 8, pre-dose: number analyzed (Participants) | 176 | 170
  GSK2167542, Week 8, pre-dose | 3237.2 (1694.66) | 3469.4 (1854.02)
  GSK2167542, Week 8, 1-3 hours: number analyzed (Participants) | 176 | 176
  GSK2167542, Week 8, 1-3 hours | 4286.3 (2514.50) | 4456.6 (2687.32)
  GSK2167542, Week 8, 4-6 hours: number analyzed (Participants) | 174 | 171
  GSK2167542, Week 8, 4-6 hours | 6238.3 (2716.05) | 6891.6 (2739.07)
  GSK2167542, Week 16 pre-dose: number analyzed (Participants) | 179 | 162
  GSK2167542, Week 16 pre-dose | 3842.4 (2428.74) | 4114.1 (2432.72)
  GSK2167542, Week 24 pre-dose: number analyzed (Participants) | 157 | 130
  GSK2167542, Week 24 pre-dose | 3617.9 (2645.51) | 4193.2 (2730.78)

7. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Analysis of absolute and relative frequencies for Adverse Event (AE) and Serious Adverse Event (SAE) by primary System Organ Class (SOC) to characterize the safety of dabrafenib and trametinib combination therapy through the monitoring of relevant clinical and laboratory safety parameters. In addition, new malignancies and AEs possibly related to study treatment were collected even if they occurred more than 30 days post-treatment. Only descriptive analysis performed.
Time Frame: From the time the first dose of study treatment administered until 30 days after discontinuation of study treatment (up to approximately 6 years).
Population: Safety Population: all randomized participants who received at least one dose of study medication and were based on the actual treatment received if this differed from that to which the participant was randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Dabrafenib + Trametinib: Crossover Dabrafenib + Trametinib
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo | Crossover Dabrafenib + Trametinib
Number analyzed (Participants) | 209 | 211 | 28
Participants
  Adverse Event (AEs) | 203 | 205 | 24
  Serious Adverse Event (SAEs) | 100 | 80 | 8

8. Post Hoc Outcome: All Collected Deaths
Description: Pre-treatment deaths were collected from screening visit up to the first day of treatment, for a maximum duration of 28 days. Patients who died during the screening period are considered as screen failure.
  On treatment deaths were collected from FPFT up to 30 days after study drug discontinuation, for a maximum duration of 77.4 months (treatment duration ranged from 0.1 to 76.4 months).
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approximately 6 years. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: up to 28 days before Day 1 (Screening), up to 77.4 months (on-treatment), up to approximately 6 years (study duration)
Population: Clinical database population; all treated patients and patients who died during screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo | Crossover Dabrafenib + Trametinib
Number analyzed (Participants) | 210 | 211 | 28
Participants
  Pre-treatment deaths | 1 | 0 | 0
  On-treatment deaths | 29 | 25 | 0
  Post-treatment deaths | 106 | 121 | 5
  All deaths | 136 | 146 | 5

ADVERSE EVENTS:
Time Frame: Adverse events were collected from First Patient First Treatment (FPFT) up to 30 days after study drug discontinuation, for a maximum duration of 77.4 months (treatment duration ranged from 0.1 to 76.4 months). In addition, new malignancies and AEs possibly related to study treatment were collected up to approximately 6 years
Description: Any clinically significant sign or symptom that occurs during the study treatment and 30 days post treatment follow up. In addition, new malignancies and AEs possibly related to study treatment were collected even if they occurred more than 30 days post-treatment.
Groups:
- All Patients: All Patients
Arm/Group | Dabrafenib + Trametinib | Dabrafenib + Placebo | Crossover Dabrafenib + Trametinib | All Patients
All-Cause Mortality (participants affected / at risk) | 135/209 | 146/211 | 5/28 | 286/420
Serious Adverse Events (participants affected / at risk) | 100/209 | 80/211 | 8/28 | 183/420
Other Adverse Events (participants affected / at risk) | 194/209 | 200/211 | 23/28 | 394/420
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib + Trametinib (N=209) | Dabrafenib + Placebo (N=211) | Crossover Dabrafenib + Trametinib (N=28) | All Patients (N=420)
Anaemia (Blood and lymphatic system disorders) | 5 | 3 | 0 | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 3 | 2 | 0 | 5
Cardiac failure (Cardiac disorders) | 0 | 2 | 1 | 3
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1
Chorioretinopathy (Eye disorders) | 1 | 1 | 0 | 2
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 1
Uveitis (Eye disorders) | 0 | 1 | 0 | 1
Visual impairment (Eye disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 0 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 3
Chest pain (General disorders) | 0 | 1 | 0 | 1
Chills (General disorders) | 10 | 3 | 0 | 13
Drowning (General disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 0 | 4
General physical health deterioration (General disorders) | 3 | 0 | 0 | 3
Influenza like illness (General disorders) | 1 | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 36 | 15 | 2 | 51
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatic haematoma (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Contrast media allergy (Immune system disorders) | 1 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1 | 0 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 6 | 2 | 0 | 8
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 1 | 0 | 2
Septic shock (Infections and infestations) | 1 | 0 | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Superinfection (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 3
Urosepsis (Infections and infestations) | 2 | 0 | 0 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural persistent drain fluid (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0 | 1 | 4
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 13 | 5 | 1 | 19
Forced expiratory volume decreased (Investigations) | 1 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1 | 0 | 1
Renal function test abnormal (Investigations) | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 1 | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Immunoglobulin G4 related disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 14 | 0 | 22
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1 | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Lipofibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Osteosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7 | 1 | 11
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 15 | 1 | 18
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 1 | 0 | 2
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 2 | 0 | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1 | 0 | 2
Facial paralysis (Nervous system disorders) | 1 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0 | 0 | 1
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 0 | 2
Syncope (Nervous system disorders) | 4 | 1 | 0 | 5
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 3 | 1 | 0 | 4
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 1 | 0 | 1
Organic brain syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 2 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 4
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 6 | 2 | 1 | 9
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib + Trametinib (N=209) | Dabrafenib + Placebo (N=211) | Crossover Dabrafenib + Trametinib (N=28) | All Patients (N=420)
Anaemia (Blood and lymphatic system disorders) | 16 | 22 | 3 | 38
Leukopenia (Blood and lymphatic system disorders) | 7 | 1 | 2 | 10
Neutropenia (Blood and lymphatic system disorders) | 20 | 5 | 3 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 2 | 2 | 13
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 2 | 6
Tachycardia (Cardiac disorders) | 6 | 13 | 3 | 21
Tinnitus (Ear and labyrinth disorders) | 5 | 2 | 3 | 9
Hypothyroidism (Endocrine disorders) | 3 | 2 | 2 | 7
Blepharitis (Eye disorders) | 2 | 0 | 2 | 4
Cataract (Eye disorders) | 2 | 4 | 3 | 8
Dry eye (Eye disorders) | 11 | 4 | 1 | 15
Vision blurred (Eye disorders) | 10 | 5 | 3 | 18
Abdominal pain (Gastrointestinal disorders) | 29 | 17 | 1 | 47
Abdominal pain upper (Gastrointestinal disorders) | 20 | 12 | 3 | 35
Constipation (Gastrointestinal disorders) | 27 | 22 | 3 | 52
Diarrhoea (Gastrointestinal disorders) | 67 | 34 | 9 | 107
Dry mouth (Gastrointestinal disorders) | 18 | 6 | 1 | 24
Nausea (Gastrointestinal disorders) | 79 | 57 | 7 | 138
Vomiting (Gastrointestinal disorders) | 57 | 31 | 3 | 89
Asthenia (General disorders) | 29 | 30 | 4 | 60
Chest pain (General disorders) | 12 | 5 | 0 | 17
Chills (General disorders) | 63 | 34 | 3 | 98
Fatigue (General disorders) | 79 | 79 | 7 | 161
Influenza like illness (General disorders) | 17 | 12 | 3 | 31
Oedema peripheral (General disorders) | 48 | 17 | 2 | 66
Pain (General disorders) | 14 | 9 | 1 | 23
Pyrexia (General disorders) | 118 | 63 | 10 | 183
Hypersensitivity (Immune system disorders) | 1 | 2 | 2 | 5
Bronchitis (Infections and infestations) | 12 | 8 | 1 | 21
Cystitis (Infections and infestations) | 11 | 2 | 0 | 13
Folliculitis (Infections and infestations) | 12 | 11 | 2 | 25
Influenza (Infections and infestations) | 17 | 7 | 5 | 28
Nasopharyngitis (Infections and infestations) | 28 | 21 | 4 | 50
Upper respiratory tract infection (Infections and infestations) | 16 | 7 | 1 | 24
Urinary tract infection (Infections and infestations) | 29 | 7 | 2 | 38
Fall (Injury, poisoning and procedural complications) | 6 | 2 | 2 | 10
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 25 | 12 | 1 | 38
Aspartate aminotransferase increased (Investigations) | 29 | 8 | 0 | 37
Blood alkaline phosphatase increased (Investigations) | 18 | 8 | 3 | 29
Blood creatine phosphokinase increased (Investigations) | 8 | 0 | 2 | 10
Blood creatinine increased (Investigations) | 8 | 2 | 2 | 12
Blood lactate dehydrogenase increased (Investigations) | 8 | 2 | 2 | 12
Ejection fraction decreased (Investigations) | 7 | 2 | 3 | 12
Gamma-glutamyltransferase increased (Investigations) | 6 | 5 | 4 | 14
Neutrophil count decreased (Investigations) | 7 | 0 | 2 | 9
Weight decreased (Investigations) | 13 | 19 | 0 | 32
Decreased appetite (Metabolism and nutrition disorders) | 30 | 28 | 5 | 60
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 1 | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 68 | 6 | 127
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 34 | 3 | 67
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19 | 7 | 3 | 29
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 4 | 2 | 11
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 14 | 11 | 0 | 25
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 19 | 1 | 31
Myalgia (Musculoskeletal and connective tissue disorders) | 27 | 28 | 3 | 56
Pain in extremity (Musculoskeletal and connective tissue disorders) | 34 | 38 | 3 | 73
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 16 | 0 | 18
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 22 | 0 | 34
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 46 | 1 | 52
Dizziness (Nervous system disorders) | 32 | 15 | 1 | 47
Dysgeusia (Nervous system disorders) | 6 | 13 | 2 | 21
Headache (Nervous system disorders) | 71 | 63 | 6 | 138
Paraesthesia (Nervous system disorders) | 9 | 12 | 1 | 22
Anxiety (Psychiatric disorders) | 12 | 6 | 3 | 21
Depression (Psychiatric disorders) | 9 | 12 | 1 | 22
Insomnia (Psychiatric disorders) | 11 | 18 | 1 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 46 | 3 | 97
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 19 | 1 | 36
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 11 | 1 | 33
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 24 | 11 | 0 | 35
Actinic keratosis (Skin and subcutaneous tissue disorders) | 12 | 15 | 1 | 27
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 61 | 0 | 80
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 21 | 8 | 0 | 29
Dry skin (Skin and subcutaneous tissue disorders) | 30 | 33 | 3 | 65
Eczema (Skin and subcutaneous tissue disorders) | 19 | 8 | 2 | 29
Erythema (Skin and subcutaneous tissue disorders) | 24 | 16 | 1 | 41
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 18 | 0 | 18
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 14 | 9 | 1 | 23
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 18 | 79 | 3 | 97
Night sweats (Skin and subcutaneous tissue disorders) | 12 | 5 | 1 | 17
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 11 | 39 | 2 | 50
Pruritus (Skin and subcutaneous tissue disorders) | 28 | 30 | 2 | 59
Rash (Skin and subcutaneous tissue disorders) | 62 | 45 | 3 | 109
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 8 | 3 | 24
Skin lesion (Skin and subcutaneous tissue disorders) | 13 | 10 | 0 | 23
Hot flush (Vascular disorders) | 8 | 5 | 2 | 15
Hypertension (Vascular disorders) | 51 | 33 | 2 | 85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.